CLINICAL TRIAL: NCT01412918
Title: Clinical Evaluation of the Inhibitor Tinnitus Treatment Masking Device & SCN9 Gene Expression
Brief Title: Inhibitor Masking Device & Sodium Channel, Voltage Gated, Type IX Alpha Subunit (SCN9) Gene Expression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of support to continue
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Marcia Dewey, AuD, Associate Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PRO00014763
Record Dates: First submitted 2011-07-06; First posted 2011-08-09 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Tinnitus
Keywords: Tinnitus; Inhibitor Device; SCN9 gene; Ringing in the ears; Milwaukee; Medical College of Wisconsin
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tinnitus (Experimental): Individual with tinnitus. Intervention: inhibitor device demonstration.
  The Inhibitor™ Tinnitus Masking Device is a new tinnitus treatment device recently available in the United States for use of temporary relief of tinnitus. The device emits an ultra high frequency sound for 60 seconds via bone conduction when applied to the mastoid. Patients reporting tinnitus will be provided the opportunity to demonstrate the device to observe any changes in their tinnitus. The device may be demonstrated up to 5 times. The investigators will be recording the the degree and duration of change in tinnitus perception following treatment with the Inhibitor™ Tinnitus Masking Device.
  Interventions: Device: The Inhibitor™ Tinnitus Masking Device
- No tinnitus (No Intervention): Individuals without tinnitus will also be masked with the device.

INTERVENTIONS:
Device: The Inhibitor™ Tinnitus Masking Device — The Inhibitor™ Tinnitus Masking Device
  Arms: Tinnitus

SUMMARY:
To evaluate the effectiveness of the Inhibitor™ Tinnitus Masking Device. To determine if there is a higher incident of expression of the sodium channel, voltage gated, type IX alpha subunit (SCN9) gene in those subjects with disturbing tinnitus than subjects that are not disturbed by tinnitus.

DETAILED DESCRIPTION:
Up to 50 million Americans have tinnitus on a regular basis with between 2-3 million suffering from tinnitus where it affects daily living. The Inhibitor™ Tinnitus Masking Device is a new tinnitus treatment device recently available in the United States for use of temporary relief of tinnitus. The device emits an ultra high frequency sound for 60 seconds via bone conduction when applied to the mastoid. Patients reporting tinnitus will be provided the opportunity to demonstrate the device to observe any changes in their tinnitus. The device may be demonstrated up to 5 times. The investigators will be recording the the degree and duration of change in tinnitus perception following treatment with the Inhibitor™ Tinnitus Masking Device. Patients may provide a genetic sample (typically via saliva sample) to look for expression of a particular genetic marker that may be associated with tinnitus. The investigators will be collect samples from both people with tinnitus and those without tinnitus to use as a control.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years,
* has tinnitus

Exclusion Criteria:

* Pacemaker,
* pregnancy,
* metal implants in head or neck,
* thrombosis, migraines/headaches,
* metal bonded retainer, surgeries within the last 6 months which patient is still recovering from,
* any medical reason your physician would advise against the use of this device,
* under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Friedland, MD, Ph.D., Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & The Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reimann F, Cox JJ, Belfer I, Diatchenko L, Zaykin DV, McHale DP, Drenth JP, Dai F, Wheeler J, Sanders F, Wood L, Wu TX, Karppinen J, Nikolajsen L, Mannikko M, Max MB, Kiselycznyk C, Poddar M, Te Morsche RH, Smith S, Gibson D, Kelempisioti A, Maixner W, Gribble FM, Woods CG. Pain perception is altered by a nucleotide polymorphism in SCN9A. Proc Natl Acad Sci U S A. 2010 Mar 16;107(11):5148-53. doi: 10.1073/pnas.0913181107. Epub 2010 Mar 8. PMID 20212137

RESULTS

PARTICIPANT FLOW:
Groups:
- Tinnitus: Individual with tinnitus.
  The Inhibitor™ Tinnitus Masking Device: The Inhibitor™ Tinnitus Masking Device
- No Tinnitus: Individuals without tinnitus.
Period: Overall Study
Arm/Group | Tinnitus | No Tinnitus
Started | 20 | 1
Completed | 20 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline participants with tinnitus demonstrating the Inhibitor™ Tinnitus Masking Device.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tinnitus | No Tinnitus | Total
Number analyzed (Participants) | 20 | 1 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 0 | 20
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 0 | 9
  Male | 11 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Determine the Percentage of Participants for Which the Inhibitor™ Tinnitus Masking Device Effected Tinnitus Perception
Description: Determine percentage of particpants with a change in tinnitus perception to evaluate the effectiveness of the Inhibitor™ Tinnitus Masking Device.
Time Frame: Single visit (day 1), assessed the day of visit
Measure: Number; unit: percentage of participants
Groups:
- Tinnitus: Tinnitus. genetic sample collection (no intervention)
Arm/Group | Tinnitus
Number analyzed (Participants) | 13
percentage of participants | 76

2. Secondary Outcome: Percentage of Participants Which Showed Presence of SCN9 Gene Expression.
Description: Percentage of participants with and without tinnitus provided a genetic sample via saliva to determine presence of SCN9 gene expression.
Time Frame: Single visit (day 1), evaluated at the time of the genetic collection.
Measure: Number; unit: % of participants with gene expression
Arm/Group | Tinnitus | No Tinnitus
Number analyzed (Participants) | 18 | 1
% of participants with gene expression | 0 | 0

ADVERSE EVENTS:
Groups:
- Tinnitus: Individual with tinnitus. Intervention: inhibitor device demonstration.
  The Inhibitor™ Tinnitus Masking Device: The Inhibitor™ Tinnitus Masking Device
Arm/Group | Tinnitus | No Tinnitus
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/1
Other Adverse Events (participants affected / at risk) | 0/20 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes